CLINICAL TRIAL: NCT05299762
Title: A Post Market Surveillance on INFUSE Bone Graft
Status: Recruiting | Type: Observational
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT21006
Record Dates: First submitted 2022-01-20; First posted 2022-03-29 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intervertebral Disc Degeneration; Spinal Fusion; Lumbar Disc Disease
Keywords: INFUSE Bone Graft; Lumbar Interbody Fusion; Anterior Lumbar Interbody Fusion; Oblique Lumbar Interbody Fusion
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients treated with the INFUSE™ Bone Graft: Patients intended to be treated with the INFUSE™ Bone Graft are eligible for enrollment. The investigator screen candidate patients against inclusion/exclusion criteria and enroll a patient only when all inclusion/exclusion criteria meet, and the patient provide written informed consent.
  Interventions: Device: INFUSE™ Bone Graft

INTERVENTIONS:
Device: INFUSE™ Bone Graft — Ministry of Food and Drug Safety (MFDS) has approved the INFUSE™ Bone Graft for anterior (ALIF) or oblique (OLIF) lumbar interbody spine fusion as a substitute for autogenous bone graft for patients with degenerative disc disease (DDD) who have had at least 6 months of non-operative treatment for this condition.

SUMMARY:
This study aims to evaluate the safety and effectiveness of INFUSE™ Bone Graft in the real-world setting in Korea.

DETAILED DESCRIPTION:
This study is a prospective, observational, multi-center, post-market surveillance to collect patient data regarding on-label use of INFUSE™ Bone Graft for lumbar fusion via ALIF or OLIF. Commercially available device will be used within its intended use.

This study is supposed to be conducted during a period of 4 years with 600 or more cases after the product approval in Korea. According to the standard of care in Korea, the patients will be followed at least 12 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Has degenerative disc disease and is indicated for lumbar interbody spine fusion from L2-S1 with INFUSE™ Bone Graft via ALIF or OLIF technique
* Agrees to participate in the study and is able to understand and sign the Informed Consent
* The procedure planned for the patient complies with the labeling of the devices that may be used in the surgical procedure
* Has at least six months of nonoperative treatment prior to the study treatment
* Is at least 18 years old at the time of informed consent

Exclusion Criteria:

* Has a known hypersensitivity to recombinant human Bone Morphogenetic Protein-2, bovine Type I collagen, or to other components of the formulation
* Has any active malignancy or undergoes treatment for a malignancy, or operative site is in the vicinity of a resected or extant tumor
* Is skeletally immature (<18 years of age or no radiographic evidence of epiphyseal closure)
* Is pregnant or lactating
* Has an active infection at the operative site or with an allergy to titanium, titanium alloy, or polyetheretherketone
* The use of the Infuse™ Bone Graft component implanted at locations other than the lower lumbar spine (e.g., cervical spine)
* Repeat applications of the Infuse™ Bone Graft component
* Has up to Grade 1 retrolisthesis
* Has hepatic or renal impairment
* Has metabolic bone disease
* Has autoimmune disease
* Has immunosuppressive disease or suppressed immune systems resulting from radiation therapy, chemotherapy, steroid therapy, or other treatments
* Is illiterate or vulnerable (e.g., the participant is incapable of judgment or is under tutelage) as per the investigator's assessment
* Concurrent participation in another clinical study that may confound study results
* Has a considerable risk for surgery
* Has a condition that could compromise study (e.g., mentally incompetent, alcohol or drug abuse) as per the investigator's assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient should be considered for enrollment if he/she is to be treated with INFUSE™ Bone Graft.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Adverse device effects by 12 months post-surgery | Surgery to 12 months
  Summarize adverse device effects
Fusion status at last assessment by 12 months post-surgery | Surgery to 12 months
  Radiographic assessment of interbody fusion will be conducted using x-rays and/or CTs

SECONDARY OUTCOMES:
Adverse events of interest up to 12 months post-surgery | Surgery to 12 months
  Summarize adverse events of interest
Clinical outcome (ODI) at 6 weeks, 3, 6, 12 months post-surgery | Baseline (pre-op) to 12 months
  Characterize changes in Oswestry Disability Index (ODI) over time. ODI evaluates how pain is affecting the patient's ability to manage in everyday life, rated on a 0 to 5 scale (higher rating represents greater disability). Improvement of ODI is defined as a decrease in score compared to baseline.
Clinical outcome (VAS) at 6 weeks, 3, 6, 12 months post-surgery | Baseline (pre-op) to 12 months
  Characterize changes in Visual Analogue Scale (VAS) for back and leg pain over time. VAS evaluates the magnitude of leg and back pain, rated on a 0 to 10 scale (higher rating represents greater pain). Improvement of VAS is defined as a decrease in score compared to baseline.
Rate of neurological success at 6 weeks, 3, 6, 12 months post-surgery | Baseline (pre-op) to 12 months
  Characterizes changes in neurological status over time. Neurological status is assessed in four sections: motor, sensory, reflexes, and straight leg raising. Following scales were used to evaluate neurological status: motor function (using 0-5 scores; 0= Total Paralysis, 1 = Palpable or Visible Contraction, 2 = Active Movement, Gravity Eliminated, 3 = Active Movement, Against Gravity, 4 = Active Movement, Against Some Resistance and 5 = Active Movement, Against Full Resistance (full strength), sensory function (using 0-2 scores; 0 = Absent, 1 = Impaired, 2 = Normal), reflexes (using 0-2 scores; 0 = Absent or Trace, 1 = Hyper-reflexic, 2 = Normal), and straight leg raise (1 = Positive, 2 = Negative).
  Overall neurological success will be defined as maintenance or improvement in all sections (motor, sensory, reflexes, and straight leg raising) for the time period evaluated (each element must remain the same or improve).

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang Gwangmyeong Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No